CLINICAL TRIAL: NCT04294186
Title: Evaluation of Factors Affecting Diaper Dermatitis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, norhan osama mohammed hassan, principle investigator, Assiut University
Other Study IDs: EOFADD
Record Dates: First submitted 2020-02-22; First posted 2020-03-03 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-03

CONDITIONS: Diaper Dermatitis
MeSH Terms: conditions — Diaper Rash

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Diaper dermatitis is one of the most common skin problems in infants and children.It is a skin disorder in the perineal , perianal and surrounding area .It frequently occurs also in areas immediately adjacent to the diaper area .

Diaper dermatitis is caused by lack of fresh air,dampness and irritation.With prevelance from 7-35 % in newborns.This skin disorder typically develops between nine and twelve months of age .

DETAILED DESCRIPTION:
The development of diaper dermatitis is multifactorial . Newborn skin exhibits a cutaneous immaturity and an increased susceptibility toward skin barrier disruption or percutaneous absorption.

The epidermal barrier function resides in the outermost epidermal layer , the stratum corneum , which is the region of terminal skin differnatiation and is composed of corneocytes . The hydrophobic components of the lipid matrix provide the epidermal permeability barrier and protect against excessive water loss and irritant penetration , whereas the corneocytes and the cornified envelope provide mechanical strength to the stratum corneum.

The skin in the diaper area is predisposed to irritation by the prolonged contact with irritants , such as urine and feces as well as by diaper occlusion, with leads to an increase in hydration and skin ph. Overhydration promotes degradation of "the brick and mortar" structure of stratum corneum, contributing to impraired barrier function.

ELIGIBILITY:
Inclusion Criteria:

* age <2 years whether male or female.
* having diaper dermatitis

Exclusion Criteria:

* age > 2 years .

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: the out patient clinic of department of dermatology,venereology and andrology , Assuit university .
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-04-18 (Estimated); Primary Completion 2020-04-18 (Estimated); Study Completion 2020-04-18 (Estimated)

PRIMARY OUTCOMES:
The percentage of patients with risk factors for Diaper dermatitis | One week
  The percentage of patients with breastfeeding, presence of diarrhea, and frequency of diaper change

REFERENCES:
- [Background] Gozen D, Caglar S, Bayraktar S, Atici F. Diaper dermatitis care of newborns human breast milk or barrier cream. J Clin Nurs. 2014 Feb;23(3-4):515-23. doi: 10.1111/jocn.12047. Epub 2013 Mar 19. PMID 23506257
- [Background] Carr AN, DeWitt T, Cork MJ, Eichenfield LF, Folster-Holst R, Hohl D, Lane AT, Paller A, Pickering L, Taieb A, Cui TY, Xu ZG, Wang X, Brink S, Niu Y, Ogle J, Odio M, Gibb RD. Diaper dermatitis prevalence and severity: Global perspective on the impact of caregiver behavior. Pediatr Dermatol. 2020 Jan;37(1):130-136. doi: 10.1111/pde.14047. Epub 2019 Dec 2. PMID 31793090
- [Background] Atherton DJ. Understanding irritant napkin dermatitis. Int J Dermatol. 2016 Jul;55 Suppl 1:7-9. doi: 10.1111/ijd.13334. PMID 27311779
- [Background] Blume-Peytavi U, Kanti V. Prevention and treatment of diaper dermatitis. Pediatr Dermatol. 2018 Mar;35 Suppl 1:s19-s23. doi: 10.1111/pde.13495. PMID 29596731
- [Result] Farahani LA, Ghobadzadeh M, Yousefi P. Comparison of the effect of human milk and topical hydrocortisone 1% on diaper dermatitis. Pediatr Dermatol. 2013 Nov-Dec;30(6):725-9. doi: 10.1111/pde.12118. Epub 2013 Apr 22. PMID 23600719
- [Result] Singalavanija S, Frieden IJ. Diaper dermatitis. Pediatr Rev. 1995 Apr;16(4):142-7. doi: 10.1542/pir.16-4-142. No abstract available. PMID 7731909